CLINICAL TRIAL: NCT07340801
Title: Analgesic Efficacy of Ultrasound-guided Inter-semispinal Fascial Plane Block (ISPB) Versus Erector Spinae Plane Block (ESPB) in Posterior Cervical Spine Surgery: A Prospective Randomized Double-Blinded Study.
Brief Title: Inter-semispinal Fascial Plane Block (ISPB) Versus Erector Spinae Plane Block (ESPB) in Posterior Cervical Spine Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mina M Fam, lecturer of Anesthesiology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R 762
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Analgesia
Keywords: the inter-semispinal fascial plane block (ISPB); the erector spinae plane (ESPB) block; Posterior cervical surgeries
MeSH Terms: conditions — Agnosia; Bites and Stings | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Active Comparator): an ultrasound-guided bilateral inter-semispinal fascial plane block (ISPB) will be performed and injection of 15 mL Bupivacaine 0.25% on each side
  Interventions: Drug: Bupivacaine
- Group (B) (Active Comparator): an ultrasound-guided bilateral erector spinae plane block (ESPB) will be performed and injection of 15 mL Bupivacaine 0.25% on each side
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — injection of 15 mL Bupivacaine 0.25% on each side

SUMMARY:
Recent advances in regional anesthesia techniques have aimed to provide more targeted and effective pain relief. Among these, the erector spinae plane (ESPB) block, the multifidus cervicis plane (MCP) block, and the paraspinal interfascial plane block (PIP) is rapidly expanding in cervical spine surgery. Of these, the inter-semispinal fascial plane block (ISPB) has gained popularity as an analgesic technique for posterior cervical spine surgery also, (ESPB) have been tried successfully for posterior cervical spine surgery in few recent trials. But to our knowledge, no study compared the efficacy of both blocks. So, the current study aimed to compare the analgesic efficacy of inter-semispinal fascial plane block versus erector spinae plane block in patients undergoing elective posterior cervical spine surgery.

DETAILED DESCRIPTION:
After approval of the institutional ethics committee, clinicaltrials.gov registration and written informed consent, (102) patients scheduled for elective Posterior Cervical Spine Surgery at Fayoum university hospital from November 2025 until the sample size is fulfilled will be enrolled in this study. This randomized double-blinded clinical trial will be reported following the tenets of the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) 2025-updated statement.

Patients will be randomized into two equal groups (1:1 allocation) using a computer-generated random number that will be sealed in a separate opaque envelope opened by an anaesthesiologist, who is responsible for performing the block and will not be involved in patient management or data collection.

For Group (A); an ultrasound-guided bilateral inter-semispinal fascial plane block (ISPB) will be performed.

For Group (B); an ultrasound-guided bilateral erector spinae plane block (ESPB) will be performed.

Inclusion criteria:

* Patients 18 years of age or older.
* Patients Scheduled for Elective Posterior Cervical Spine Surgery.
* American Society of Anesthesiologists (ASA) physical status I-III.

Exclusion criteria:

* Patients with traumatic or emergency surgeries.
* Renal or hepatic impairment
* Allergy to drug used.
* Re-do surgery.
* Coagulopathy.
* Neuromuscular disease.
* Preoperative poor left ventricular function (EF < 35%).
* Systemic infections or infections at site of injection.
* Psychiatric illnesses (schizophrenia, bipolar, uncontrolled anxiety or depression).
* Narcotic dependency.

ANESTHETIC TECHNIQUE:

Anesthesia and Perioperative Management:

After taking a complete history, all patients will be preoperatively examined and routinely investigated with complete blood count, coagulation profile, hepatic, renal functions, electrolytes and arterial blood gases as well, Chest-x ray and echocardiography will be requested on demand. Before the induction of anesthesia, 18G cannula will be inserted for venous access. Standard ASA monitoring, including non-invasive blood pressure (NIBP), heart rate (HR), peripheral oxygen saturation (SpO2), and electrocardiogram (ECG) monitoring, will be performed continuously throughout the procedure. After pre-oxygenation, anesthesia induction will be carried out with the following medication: Fentanyl 1 μg/kg IV, Propofol 2 mg/kg IV and atracurium 0.5 mg/kg IV. Once adequate muscle relaxation is achieved, endotracheal intubation will be performed using a cuffed endotracheal tube, and patients will be placed prone on bolsters with the neck in neutral alignment, ensuring all pressure points are padded. Anesthesia will be maintained with a mixture of 50% O2, 50% medical air, and 1.2% isoflurane, along with 0.5 mg/kg atracurium for maintenance dosing as required. Mechanical ventilation will be adjusted to maintain normocapnia.

After induction of anesthesia and adequate positioning of the patient; the solution for the block will be prepared and the US machine will be turned on, the skin on either side of the incision will be prepared with povidone iodine solution then, all attendees will leave the OR apart from an anaesthesiologist who will perform the block according to the randomization number and a trained nurse for assistance. During this time patient monitoring will be the responsibility of that team and reported automatically via the OR monitors.

For inter-semispinal fascial plane block:

A linear ultrasound probe 2-5 MHz (Philips clear vue350, Philips healthcare, Andover MAO1810, USA, Machine ID: 1385, Nile medical centre, service@nilemed.net) will be used. Linear probe orientation in the transverse plane will be used to identify the five-layered posterior cervical muscles at the level of C5. By sliding the probe cranially, we will able to count the fifth cervical spine from the C7 spinous process. A 23 G 90 mm Quincke's spinal needle (B Braun, Melsungen, Germany) is inserted in-plane through the skin and advanced into the fascial plane between the semispinalis cervicis and semispinalis capitis muscles under continuous ultrasound guidance. The correct needle tip position under the semispinalis capitis is confirmed by hydro-dissection using 1 mL of normal saline, followed by injection of 15 mL Bupivacaine 0.25%. Correct drug placement will be confirmed by the linear spread of the local anaesthetic drug, which separates the semispinalis capitis and semispinalis cervicis muscles. The spread of the drugs proximally and distally is confirmed through ultrasound. A similar mixture will be administered on the other side too.

The erector spinae plane block:

For performing the block, a 2-5 MHz linear probe will be used to identify the T1 vertebral level. Once the T1 vertebral level identified, the probe will be moved in a longitudinal parasagittal orientation 3 to 4 cm lateral to the midline to identify the tip of the transverse process of T1. A 23G 90 mm Quincke's spinal needle (B Braun, Melsungen, Germany) will be inserted from a caudo-cranial angulation to contact the T1 transverse process. Correct needle tip position under the erector spinae will be confirmed by hydro dissection using 1 ml of Normal Saline followed by injection of 15 ml Bupivacaine 0.25%. Correct drug placement will be confirmed by the linear spread of the local anesthetic drug separating the erector spinae muscle from the transverse processes. The spread of the drugs proximally into the sub-axial cervical spine will be confirmed through ultrasound. The same technique will be repeated for the other side.

After performing the block the investigators, data collectors and the surgeons will enter the OR, and the surgery will be performed. During surgery, a rescue fentanyl will be given with a dose of 0.5µg/kg when needed guided by the Surgical Pleth Index (SPI). Blood pressure and heart rate will be continuously monitored. Hypotension (SBP <90 mmHg or ≥20% below baseline) will be managed with 5 mg IV ephedrine; bradycardia (HR ≤50 bpm) will be managed with 0.5 mg IV atropine.

By end of surgery, IV neostigmine and atropine will be used to reverse residual neuromuscular blockade. Patients will be extubated upon full recovery and transferred to the post-anesthesia care unit (PACU), and subsequently to the ward when a modified Aldrete score ≥9 was achieved.

Management of Postoperative Pain During the preoperative consultation, all patients will be instructed on the utilization of the PCA device and the 11-point NRS (0 = no pain, 10 = worst pain). Postoperative pain will be assessed at 0, 6, 12, 18, and 24 hours post-surgery by an investigator blinded to group allocation.

Postoperative analgesia will include IV paracetamol 1 g every 8 hours, based on the routine hospital protocol. Additional analgesia will be provided using a PCA device delivering IV fentanyl (conc. 10 μg.ml-1) with bolus of 15 μg, and lockout interval 10 minutes, maximum cumulative dose of 90μ.hr-1 and no background dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Patients Scheduled for Elective Posterior Cervical Spine Surgery.
* American Society of Anesthesiologists (ASA) physical status I-III.

Exclusion criteria:

* Patients with traumatic or emergency surgeries.
* Renal or hepatic impairment
* Allergy to drug used.
* Re-do surgery.
* Coagulopathy.
* Neuromuscular disease.
* Preoperative poor left ventricular function (EF < 35%).
* Systemic infections or infections at site of injection.
* Psychiatric illnesses (schizophrenia, bipolar, uncontrolled anxiety or depression).
* Narcotic dependency.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The total perioperative opioid consumption | during the first 24 hours postoperatively
  the total perioperative opioid consumption through two co-primary outcomes, i.e. total amount of fentanyl administered intraoperatively and total fentanyl consumption during the first 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mahdy Abdelhady, MD, Principal Investigator — Fayoum University
Locations (1):
- Fayoum University Hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmoud AM, Alsaied MA, Ragab SG, Abdelfattah YA, Farghaly OS, Shawky MA. Inter-Semispinalis Plane Block Versus General Anesthesia for Postoperative Analgesia in Posterior Cervical Spine Surgery: A Randomized Controlled Trial. Anesth Pain Med. 2024 Feb 16;14(1):e143369. doi: 10.5812/aapm-143369. eCollection 2024 Feb. PMID 38725919
- [Background] Abdelhaleem NF, Youssef EM, Hegab AS. Analgesic efficacy of inter-semispinal fascial plane block in Patients undergoing Cervical Spine Surgery through Posterior Approach: a randomized controlled trial. Anaesth Crit Care Pain Med. 2023 Aug;42(4):101213. doi: 10.1016/j.accpm.2023.101213. Epub 2023 Mar 7. PMID 36894055